CLINICAL TRIAL: NCT01270997
Title: A Multicenter Randomized Double-blind Active-controlled Parallel Group Phase Ⅲ Trial to Evaluate the Equivalence in Efficacy and Safety of HD203 and Enbrel in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: Randomized Double-blind Parallel Trial to Evaluate Equivalence in Efficacy and Safety of HD203 and Enbrel in RA Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanwha Chemical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAGLE-III-10
Record Dates: First submitted 2011-01-02; First posted 2011-01-06 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD203 (Experimental): Subcutaneous injection (SC) HD203 25mg twice a week for 48 weeks
  Interventions: Biological: Etanercept
- Enbrel (Active Comparator): Subcutaneous injection (SC) Enbrel® 25mg twice a week for 48 weeks.
  Interventions: Biological: Etanercept

INTERVENTIONS:
Biological: Etanercept — Subcutaneous injection (SC) Etanercept 25mg twice a week for 48 weeks
  Other Names: HD203
  Arms: HD203
Biological: Etanercept — Subcutaneous injection (SC) Etanercept 25mg twice a week for 48 weeks
  Other Names: Enbrel
  Arms: Enbrel

SUMMARY:
The objective is to prove the equivalence in efficacy and safety of HD203 and Enbrel® in combination with Methotrexate in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Primary Objective:

To prove the equivalence between two groups by comparing the ACR20 of W24 with the baseline after injecting HD203 25mg and (Enbrel®) 25mg into the patients with rheumatoid arthritis for 24 weeks.

Secondary Objective:

To compare the efficacy of ACR20, ACR50 and ACR70, etc along with safety in adverse event, vital signs, Laboratory test, physical examination and immunogenicity, etc between two groups with baseline after injecting HD203 25mg and (Enbrel®) 25mg into patients with rheumatoid arthritis for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are 20 or over
* Patients who satisfy the classification criteria of Rheumatoid Arthritis according to American Colleague of Rheumatology (ACR 1987)
* Patients who are applicable to functional status I - III of American Colleague of Rheumatology

Exclusion Criteria:

* Patients who have autoimmune diseases other than rheumatoid arthritis or have significant secondary systematic disease caused by rheumatoid arthritis
* Patients who are currently participating in other clinical studies or receiving treatment for drugs not sold in the market or for experiment
* Patients who have significant other diseases that may affect the clinical trial when judged by the clinical trial Investigator
* In the opinion of the investigator, may put the patient at risk because of participation on the study or may influence the patients' ability to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To prove the equivalence between two groups by comparing the ACR20 of W24 with the baseline after injecting HD203 and Enbrel® into rheumatoid arthritis patients for 24 weeks. | 24week

SECONDARY OUTCOMES:
To compare the efficacy of ACR20, ACR50 and ACR70 along with safety and immunogenicity between two groups with baseline after injecting HD203 and Enbrel® into rheumatoid arthritis patients for 48 weeks | 12W, 24W, 48W

CONTACTS AND LOCATIONS:
Overall Officials: Sang Chul Bae, MD, PhD, MPH, Principal Investigator — Hanyang University College of Medicine
Locations (1):
- Hospetal for Rheumatic Diseases Hanyang University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Bae SC, Kim J, Choe JY, Park W, Lee SH, Park YB, Shim SC, Lee SS, Sung YK, Choi CB, Lee SR, Park H, Ahn Y; HERA Study Investigators. A phase III, multicentre, randomised, double-blind, active-controlled, parallel-group trial comparing safety and efficacy of HD203, with innovator etanercept, in combination with methotrexate, in patients with rheumatoid arthritis: the HERA study. Ann Rheum Dis. 2017 Jan;76(1):65-71. doi: 10.1136/annrheumdis-2015-207613. Epub 2016 Feb 23. PMID 26905864